CLINICAL TRIAL: NCT04510246
Title: A Randomised Controlled Trial of Active Case Management to Link Hepatitis C Notifications to Hepatitis C Treatment in Tasmania
Brief Title: Link Hepatitis C Notifications to Treatment in Tasmania
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tas RCT HCV Notifications
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: This study will be a two-armed cluster randomised controlled trial with randomisation at the level of the general practitioner.
Who Masked: Participant, Investigator
Masking Description: Given the nature of the intervention, it is impossible to blind either the health care worker or the general practitioner to allocation. However, the analysis will be conducted by an analyst at the Burnet Institute who will not have contact with the general practitioners and will be blinded to intervention allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Practitioners randomised to the intervention arm will receive the standard of care surveillance letter if the notification is new. Both new and repeat notifications will receive further enhanced case support during the project if required. Support can be provided at the first phone call, or if accepted and required, in a 12-week period during which the DoH health care worker can do follow-up calls with the GP or directly with the patient to inform the patient and enhance linkage back to their GP. At the end of the 12-week period, a follow-up call we be carried out for the project evaluation.
  Interventions: Behavioral: Enhanced case management
- Control (No Intervention): All practitioners randomised to this arm will be contacted by telephone approximately 12 weeks after an HCV notification has been made from the laboratory to the Department of Health.This is not current standard practise and will be performed by the DoH HCV health worker for the project evaluation purpose. At this phone call consent will be sought for the GP to provide information on their clinical management of the notified patient. The details of the clinical management survey are provided as Appendix B. Details provided or missing from the standard DoH surveillance form would be confirmed with the GP at this phone call. Three attempts will be made to contact the practitioner to complete the survey within a 30-day period before they are determined to be unable to be contacted.

INTERVENTIONS:
Behavioral: Enhanced case management — The health care worker will offer support to the GP for all aspects of the cascade of hepatitis C care including:
  * Further testing advice
  * Awareness that treatment can be prescribed by the general practitioner
  * Conducting pre-treatment work-up assessment
  * DAA prescription guidelines, including linkage to specialist consultation
  * Providing treatment support
  * Advising on testing process for cure
  * Advising on post-cure management including methods of follow-up to manage risks (e.g. harm minimisation, reducing re-infection risk, opioid substitution therapy)
  * Linking GP to resources for patients with cirrhosis or other concerns to specialist support for ongoing management.
  The GP will be offered the option of the DoH specialist to contact the patient directly with the GP's consent to notify them of their result and to educate them on testing and treatment options and referral back to their GP.
  Arms: Intervention

SUMMARY:
This project will utilise the notification process as a point of intervention to work with primary practitioners (GP) by contacting them directly when a notification of hepatitis C exposure is received by the Tasmanian department of Health (DoH). A designated role will exist within DoH of a specialist HCV health worker to contact GPs to provide supported assistance in the process of the follow up hepatitis C diagnoses with patients. The study will evaluate whether active follow up of providers with enhanced case management is effective in having patients linked to hepatitis C treatment compared to current standard of care of surveillance for new notifications. The study will also compare the cost-effectiveness of this approach compared to current standard of care after one of their patients is notified with a positive hepatitis C antibody result.

ELIGIBILITY:
Inclusion Criteria:

* General Practitioners (GP) who have requested a hepatitis C test that leads to new or repeat notification to the Tasmanian Department of Health

Exclusion Criteria:

* Not based in Tasmania
* Practitioner from correctional service
* Specialist
* Nurse practitioner who initiated test
* Sexual health service doctor
* Family planning
* Trainee

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases notified with hepatitis C who commence hepatitis C treatment | The study follow up period is 12 weeks
  The primary outcome will be the proportion of cases notified with hepatitis C who commence hepatitis C treatment within 12 weeks of initial contact. This will be assessed using the information provided by practitioners at the 12-week follow-up phone call and will be compared across the two arms.

SECONDARY OUTCOMES:
Proportion of people diagnosed with hepatitis C with a documented HCV RNA test result | The study follow up period is 12 weeks
  The the proportion of cases notified with hepatitis C with documented HCV RNA results within 12 weeks of initial contact. This will be assessed using lab data and information provided by practitioners.
Proportion of people diagnosed with hepatitis C completing treatment work-up blood tests | The study follow up period is 12 weeks
  The the proportion of HCV RNA positive cases who completed treatment work up blood tests within 12 weeks of initial contact. This will be assessed using lab data and information provided by practitioners.
Proportion of people diagnosed with hepatitis C completing an appropriate course of hepatitis C treatment as prescribed | The study follow up period is 12 weeks
  The the proportion of HCV cases who complete an appropriate course of prescribed hepatitis C treatment..

CONTACTS AND LOCATIONS:
Locations (1):
- Tasmanian Department of Health, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data will be captured in RedCap and is de-identifiable and will be shared as a data file from the data capturing tool.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of study completion
Access Criteria: Full data file will be available to be shared after study completion.

REFERENCES:
- [Derived] Marukutira T, Moore KP, Hellard M, Richmond J, Turner K, Pedrana AE, Melody S, Johnston FH, Owen L, Van Den Boom W, Scott N, Thompson A, Iser D, Spelman T, Veitch M, Stoove MA, Doyle J. Randomised controlled trial of active case management to link hepatitis C notifications to treatment in Tasmania, Australia: a study protocol. BMJ Open. 2022 Mar 25;12(3):e056120. doi: 10.1136/bmjopen-2021-056120. PMID 35338062